CLINICAL TRIAL: NCT04871425
Title: Ketamine Versus Fentanyl for Surgical Abortions: A Randomized Controlled Noninferiority Trial
Brief Title: Ketamine Versus Fentanyl for Surgical Abortions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Jennifer Chin, Fellow, Family Planning: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00012218
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Abortion in First Trimester; Pain, Procedural; Opioid Use
MeSH Terms: conditions — Pain, Procedural | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participant will receive 2mg IV midazolam and 0.2-0.5mg/kg IV ketamine over 2 minutes, which can be repeated q5 minutes until appropriate analgesia is achieved.
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): Participant will receive 2mg IV midazolam and 0.5-1mcg/kg IV fentanyl over 2 minutes, which can be repeated q5m until appropriate analgesia is achieved.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — IV ketamine
  Arms: Ketamine
Drug: Fentanyl — IV fentanyl
  Arms: Fentanyl

SUMMARY:
Ketamine is commonly used for procedural sedation and analgesia. It is widely used for trauma cases in the emergency department and is considered a superior agent in the outpatient setting due to its lack of respiratory and cardiovascular depression. In chronic opioid users, ketamine decreases acute pain and reduces postoperative opioid consumption. Few studies have examined the use of ketamine for surgical abortions. Previous studies found significant rates of emergence phenomena; however, this can be prevented if a benzodiazepine is given at the same time. Ketamine deserves further study to determine whether it is an acceptable alternative to a standard opioid-based regimen for surgical abortion. Our primary objective is to compare patient satisfaction after surgical abortion among patients receiving IV ketamine versus IV fentanyl for procedural sedation. Our secondary objectives include postoperative pain, additional pain medication used, and postoperative opioid use after the procedure. Our hypothesis is that ketamine will provide similar patient satisfaction and reduce postoperative opioid use. This will be a randomized controlled noninferiority clinical trial of 84 women receiving either IV ketamine with IV midazolam or IV fentanyl with IV midazolam for outpatient one day surgical abortions up to 13, 6/7 weeks gestation. Both groups will receive a standardized paracervical block and additional pain medication as needed. Our study has the potential to introduce IV ketamine as a satisfactory medication for outpatient surgical abortions. Ketamine may decrease the need for IV fentanyl, reduce postoperative opioid use, and may prove to be a superior analgesic for chronic opioid users.

DETAILED DESCRIPTION:
First-trimester surgical abortions are one of the most common outpatient procedures worldwide. Although abortion is a quick procedure, most patients still report at least moderate pain.1 Most providers use a paracervical block plus intravenous (IV) moderate sedation with fentanyl (38%) or oral medication (33%). A recent trial comparing IV fentanyl to placebo among participants who also received the paracervical block found a 1-point difference in pain on an 11-point scale. The authors questioned the benefit of this reduction in pain in light of fentanyl's various side effects including nausea and drowsiness, the requirement for additional monitoring and resuscitative equipment, and need for naloxone in case of overdose.

Due to our nation's opioid crisis, there has been growing interest in identifying a non-opioid medication to provide safe, short term, satisfactory pain control during first trimester outpatient surgical abortions. Ketamine is commonly used for procedural sedation and analgesia, and it also reduces postoperative pain. It acts primarily as an N-methyl-D-aspartate receptor antagonist but has some opioid receptor activity. It is widely used for trauma cases and acute pain crises, and is considered a superior agent in the outpatient setting due to its lack of respiratory and cardiovascular depression. Few studies have examined ketamine for surgical abortions. Most studies found improvement when compared to the paracervical block or remifentanil. Our study's primary outcome was to determine if ketamine was noninferior in terms of patient satisfaction with anesthesia to fentanyl for procedural sedation for outpatient first trimester surgical abortions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 years or older
* Voluntarily requesting surgical pregnancy termination
* Intrauterine pregnancy up to 13 weeks 6 days by transabdominal or transvaginal ultrasound performed on day of procedure
* Eligible for suction curettage
* English or Spanish speaking
* Able and willing to give informed consent and agree to terms of the study

Exclusion Criteria:

* Age less than 14 years
* Reaspiration procedure or failed medication abortion
* Early pregnancy loss
* Alcohol use disorder or acute alcohol intoxication
* Currently incarcerated
* Gestational age 14 weeks or more
* Requesting a specific pain regimen
* Premedication with misoprostol
* Contraindications or allergies to ketamine or fentanyl

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chin, MD, Principal Investigator — Fellow
Locations (1):
- Cedar River Clinic, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chin J, McGrath M, Lokken E, Upegui CD, Prager S, Micks E. Ketamine Compared With Fentanyl for Surgical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2022 Sep 1;140(3):461-469. doi: 10.1097/AOG.0000000000004903. Epub 2022 Aug 3. PMID 35926204

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Fentanyl
Started | 57 | 53
Completed | 42 | 45
Not Completed | 15 | 8

BASELINE CHARACTERISTICS:
Population: We recruited and randomized 110 participants. After randomization, five participants in the ketamine group were excluded due to two participants receiving the wrong medication, one participant not achieving IV access, one not having transportation, and one being hypertensive. Thus, 52 participants received ketamine and 53 participants received fentanyl.
Groups:
- Fentanyl: Participant will receive 2mg IV midazolam and 0.2-0.5mg/kg IV fentanyl over 2 minutes, which can be repeated q5 minutes until appropriate analgesia is achieved.
  Fentanyl: IV fentanyl
- Ketamine: Participant will receive 2mg IV midazolam and 0.5-1mcg/kg IV ketamine over 2 minutes, which can be repeated q5m until appropriate analgesia is achieved.
  Ketamine: IV ketamine
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Ketamine | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.4) | 27.6 (5.8) | 27.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 105
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 43 | 42 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 7 | 21
  White | 17 | 24 | 41
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 11 | 13 | 24
Gestational age [Mean (Standard Deviation); unit: weeks] | 6.4 (1.8) | 7.4 (2.3) | 6.7 (2)

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Anesthesia Assessed by the ISAS
Description: After the procedure, either at time of discharge (if less than 30 minutes) or at 30 minutes (if not yet discharged), research personnel will assess the participant's satisfaction with anesthesia using the Iowa Satisfaction with Anesthesia Scale. This is a validated perioperative anesthesia satisfaction scale with a minimum score of -3 and a maximum score of +3 with higher scores indicating higher satisfaction.
Time Frame: At discharge or 30 minutes after the procedure
Population: We randomized 110 participants: 57 in the ketamine group and 53 in the fentanyl group. After randomization, an additional five participants in the ketamine group were excluded due to two participants receiving the wrong medication, one participant not achieving IV access, one not having transportation, and one being hypertensive. Thus, 52 participants received ketamine and 53 participants received fentanyl.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 52 | 53
score on a scale | 2.4 (0.8) | 2.2 (0.9)

2. Secondary Outcome: Provider Satisfaction With Anesthesia Assessed by the VAS
Description: After the procedure, research personnel will assess provider's satisfaction with patient's anesthesia on a 100mm visual analog scale. The minimum score is 0mm and the maximum score if 100mm, with higher scores indicating higher satisfaction.
Time Frame: Immediately postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 52 | 53
score on a scale | 90 (15.8) | 86.8 (21.3)

3. Secondary Outcome: Number of Participants Administered Additional Pain Medications
Description: After the procedure, research personnel will ask anesthetist what medications, if any, they gave outside of the study protocol
Time Frame: Immediately postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 52 | 53
Participants | 23 | 30

4. Secondary Outcome: Postoperative Pain Assessed by the VAS
Description: Patients will complete 2 followup surveys asking about their postoperative pain after discharge. This will be assessed on a 100mm visual analog scale. The minimum score is 0mm and the maximum score if 100mm, with higher scores indicating higher pain levels.
Time Frame: 24 hours postoperatively and 7 days postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Fentanyl
Number analyzed (Participants) | 52 | 53
score on a scale
  Pain post-op day 1 | 24.5 (24.2) | 22 (23)
  Pain post-op day 7 | 18.2 (21) | 19.1 (27.1)

ADVERSE EVENTS:
Time Frame: 1 week after procedure
Description: We randomized 110 participants: 57 in the ketamine group and 53 in the fentanyl group. After randomization, an additional five participants in the ketamine group were excluded due to two participants receiving the wrong medication, one participant not achieving IV access, one not having transportation, and one being hypertensive. Thus, 52 participants received ketamine and 53 participants received fentanyl.
Arm/Group | Ketamine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT04871425/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT04871425/ICF_001.pdf